CLINICAL TRIAL: NCT03426475
Title: Effects of Strategies to Improve General Practitioner-nurse Collaboration and Communication in Regard to Hospital Admissions of Nursing Home Residents.
Brief Title: Effect of Strategies to Improve General Practitioner-nurse Collaboration and Communication
Acronym: interprof ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Karsten Gavenis, Clinical Study Management on behalf of the Principal Investigator, University Medical Center Goettingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01811
Record Dates: First submitted 2017-12-05; First posted 2018-02-08 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Utilization of Medical Care by Nursing Home Residents
Keywords: nursing home residents; interprofessional collaboration; reduction of hospitalisation

STUDY DESIGN:
Masking Description: Blinded study nurses with respect of primary outcome.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Care of nursing home residents as usual.
- Interventional Group (Experimental): Implementation of interprof ACT measures to improve collaboration and communication between general practitioners and nursing staff. Measures are selected and adapted by nursing home management / nurses, GPs and residents' relatives or representatives.
  Interventions: Procedure: interprof ACT measures

INTERVENTIONS:
Procedure: interprof ACT measures — Definition of common goals between general practitioner and nursing staff, appointment of a contact person, support in assigning medication, use of name badges worn by GPs and nurses during visits, mandatory availability of contact person, standardized procedures for GPs home visits
  Arms: Interventional Group

SUMMARY:
Previously,six measures were developed for a better collaboration of general practitioners and nurses in nursing homes in a qualitative multistep bottom-up process. These measures, summarised as the interprof ACT intervention, shall improve the flow of information and the communication between the involved parties and lead to more transparency and effectiveness regarding treatment decisions of nursing home residents.The major aim of this trial is to examine the clinical effectiveness of interprof ACT. The main hypothesis is that implementation of interprof ACT reduces the cumulative incidence of hospitalisations of nursing home residents within 12 months from 50% to 35% (15% absolute reduction).

ELIGIBILITY:
Inclusion Criteria Residents:

* at least one GP visit in recent three months or
* two GP visits in recent 6 months or
* admission to the nursing home during the precedent 6 months independently of documented GP contacts
* at least 18 years of age
* written informed consent by the resident or her/his legal guardian

Inclusion Criteria Nursing Homes:

* minimum size of 40 residents
* written consent provided by the nursing home Manager Prior to randomisation

Exclusion Criteria Residents:

- admission for short term care only

Exclusion Criteria Nursing Homes:

- participation in other projects on interprofessional collaboration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
cumulative number of hospitalisation | within 12 months
  Cumulative incidence of hospitalisations from nursing home residents within 12 months

SECONDARY OUTCOMES:
absolute number of hospitalisations | within 12 months
  number of hospitalisations within 12 months
hospital days | within 12 months
  Hospital days within 12 months
mortality | within 12 months
  mortality within 12 months
potentially inadequate medications | baseline and after 6 and 12 months
  potentially inadequate medications at baseline and for follow-ups at 6 and 12 months
Adverse Events | within 12 months
  Adverse Events within 12 months
Quality of Life in Alzheimer's Disease scale - Nursing Home version (QoL-AD-NH) | baseline and after 12 months
  Residents' quality of life at baseline and at 12 months. Scale range is 15 - 60, with higher scores indicating higher QoL.
Health-related Quality of Life (HRQL) of residents measured by EQ-5D-5L | baseline and after 12 months
  The EQ-5D-5L consist of two self-rating components: the EQ-5D descriptive system and a visual analogue scale (EQ VAS). The EQ-5D descriptive system measures HRQL on the five dimensions "mobility", "self-care", "usual activities", "pain / discomfort" and "anxiety / depression". On each dimension participants can rate either "no problems" (0), "slight problems" (1), "moderate problems" (2), "severe problems" (3) or "extreme problems" (4), resulting in a score ranging from 0 (best) to 4 (worst). The scores of the single dimensions can be combined to a sum score ranging from 0 (best) to 20 (worst). In addition, so called "utility weights" can be attached to any possible combination of answers on the EQ-5D descriptive system which results in a utility score ranging from 0 (death) to 1 (full HRQL), which is then used to calculate quality-adjusted life years (QALYs). The EQ VAS ranges from 0 (worst imaginable health state) to 100 (best imaginable health state).
medical services | within 12 months
  use of other medical services within 12 months
economic evaluation: efficiency | after 12 months
  economic evaluation: efficiency (incremental cost-effectiveness ratio) and cost savings from payer and societal perspective
Quality of inter-professional collaboration according to the Partnership Self-Assessment Tool (PSAT) score | after 12 months
  Higher score values indicating better collaboration.
Attitudes towards inter-professional collaboration according to the Jefferson Scale of Attitudes Toward Physician-Nurse Collaboration (JSAPNC) score | after 12 months
  Higher score values indicating more favourable attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Hummers, Prof. Dr. med., Principal Investigator — Department of General Practice, University Medical Center Goettingen
Locations (4):
- Germany (4):
  - Department of General Practice, University Medical Center Göttingen, Göttingen
  - Organization and Corporate Development, Georg August University Göttingen, Göttingen
  - Department of General Practice/Primary Care, University Medical Center Hamburg-Eppendorf, Hamburg
  - Institute for Social Medicine and Epidemiology, Nursing Research Group,University of Lübeck, Lübeck

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazur A, Tetzlaff B, Mallon T, Hesjedal-Streller B, Wei V, Scherer M, Kopke S, Balzer K, Steyer L, Friede T, Pfeiffer S, Hummers E, Muller C. Cluster randomised trial of a complex interprofessional intervention (interprof ACT) to reduce hospital admission of nursing home residents. Age Ageing. 2023 Mar 1;52(3):afad022. doi: 10.1093/ageing/afad022. PMID 36934341
- [Derived] Steyer L, Kortkamp C, Muller C, Tetzlaff B, Fleischmann N, Weber CE, Scherer M, Kuhn A, Jarchow AM, Luth F, Kopke S, Friede T, Konig HH, Hummers E, Maurer I, Balzer K. Implementation, mechanisms of change and contextual factors of a complex intervention to improve interprofessional collaboration and the quality of medical care for nursing home residents: study protocol of the process evaluation of the interprof ACT intervention package. Trials. 2022 Jul 8;23(1):561. doi: 10.1186/s13063-022-06476-6. PMID 35804455
- [Derived] Muller C, Hesjedal-Streller B, Fleischmann N, Tetzlaff B, Mallon T, Scherer M, Kopke S, Balzer K, Gartner L, Maurer I, Friede T, Konig HH, Hummers E. Effects of strategies to improve general practitioner-nurse collaboration and communication in regard to hospital admissions of nursing home residents (interprof ACT): study protocol for a cluster randomised controlled trial. Trials. 2020 Nov 5;21(1):913. doi: 10.1186/s13063-020-04736-x. PMID 33153484